CLINICAL TRIAL: NCT02295332
Title: A Study of RG7625 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: WP29542; 2014-003538-23 (EudraCT Number)
Record Dates: First submitted 2014-11-17; First posted 2014-11-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Cohort A (Experimental)
  Interventions: Drug: Placebo; Drug: RG7625
- Cohort B (Experimental)
  Interventions: Drug: Placebo; Drug: RG7625

INTERVENTIONS:
Drug: Placebo — Matching oral placebo capsules to RG7625, according to treatment schedule
Drug: RG7625 — oral administration, capsules, single ascending dose according to treatment schedule

SUMMARY:
This is a single center, randomized, double-blind, placebo-controlled, single ascending dose study that will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamic effects of single doses of RG7625 in healthy male and female volunteers.

The study will employ an interleaved cohort ('leapfrog') design in which dosing is alternated between two cohorts and each individual within a cohort will receive study drug dosing on four occasions - in effect giving a four treatment, four period, four-way crossover for each individual. The minimum duration for each participant is approximately 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants, 18 to 60 years of age, inclusive
* A body mass index between 18 to 30 kg/m2 inclusive
* Able to participate and willing to give written informed consent and to comply with the study restrictions

Exclusion Criteria:

* Any clinically relevant abnormalities, concomitant diseases or ongoing medical conditions, abnormal laboratory test results or a history of any other clinically significant disorders
* Any major illness within the one month preceding the screening visit, or any febrile illness within the two weeks preceding the screening visit
* Any significant allergic reaction to drugs
* Immunocompromised or with reduced immune function and/or immunization within 30 days before the first study drug administration or planning vaccination during the study
* Women who are pregnant or lactating or of childbearing potential
* Clinically significant abnormal ECG or other risk factors for QT prolongation
* Use of prescribed or over the counter medication
* Inability or unwillingness to comply with study requirements

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2014-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Safety (composite outcome measure):Incidence and severity of adverse events (AEs), laboratory abnormalities, changes in ECG, vital signs | Approximately 22 weeks

SECONDARY OUTCOMES:
Pharmacokinetics (composite outcome measure): PK profile and parameters derived from plasma concentrations of RG7625 and its metabolites [AUCinf, AUClast, Cmax, tmax, t1/2, CL/F, V/F, Ae, fe and CLR] | 22 weeks
Pharmacodynamics (composite outcome measure): measurement of intracellular p10 concentrations and cell surface expression of major histocompatibility complex class (MHC)-II, relationship to RG7625 exposure | 22 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Zuidlaren, Netherlands

REFERENCES:
- [Derived] Theron M, Bentley D, Nagel S, Manchester M, Gerg M, Schindler T, Silva A, Ecabert B, Teixeira P, Perret C, Reis B. Pharmacodynamic Monitoring of RO5459072, a Small Molecule Inhibitor of Cathepsin S. Front Immunol. 2017 Jul 17;8:806. doi: 10.3389/fimmu.2017.00806. eCollection 2017. PMID 28769925